CLINICAL TRIAL: NCT02633592
Title: Seated Evaluation of Anorectal funcTion by High Resolution Anorectal Manometry: a Randomized Comparison of Measurements in the Seated and Left Lateral Positions
Brief Title: Seated Evaluation of Anorectal funcTion by High Resolution Anorectal Manometry
Acronym: SEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KEK-ZH-Nr. 2014-0058
Record Dates: First submitted 2015-11-27; First posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Anismus; Incontinence
Keywords: High Resolution Anorectal Manometry; Magnetic Resonance Imaging; Balloon Expulsion; Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HRARM (Active Comparator): Patients and healthy volunteers are subjected to position change ( LLP to SP) during pressure measurements with HR-ARM.
  Interventions: Other: HRARM
- MRI Defecography (Active Comparator): Patients and healthy volunteers are subjected to position change during MRI Defecography
  Interventions: Other: MRI Defecography

INTERVENTIONS:
Other: HRARM — Patients and healthy volunteers are investigated in the seated and lying position during HRAM
  Arms: HRARM
Other: MRI Defecography — Patients and healthy volunteers are investigated in the supine and left lateral position in the MRI
  Other Names: MRD
  Arms: MRI Defecography

SUMMARY:
To assess whether HR-ARM (High resolution Anorectal Manometry) performed in the more naturalistic / physiological upright, seated position on a commode provides a more valid assessment of anorectal function and simulated defecation than the same test performed in the standard, left lateral position

DETAILED DESCRIPTION:
High Resolution Anorectal Manometry (HR-ARM) with data presented as pressure topography is a recent addition to the tests available for diagnosis of defecatory disorders including fecal incontinence and constipation.HR-ARM represents an advance on conventional manometry because closely spaced sensors across the anal sphincter remove the need for a pull-through procedure and facilitate data acquisition and interpretation. In particular measurements are not confounded by changes in position of the catheter relative to anal sphincter that occur during voluntary contraction and, especially, simulated defecation.

Notwithstanding these technological improvements, important concerns remain about the validity of manometry measurements during simulated defecation. These concerns are based on the observation in both conventional and HR-ARM that a large proportion of healthy individuals appear to have abnormal anorectal function ("dyssynergia") during simulated defecation.This limitation led to the recommendation that the finding of dyssynergia on manometry should be confirmed by defecography. This is unsatisfactory as diagnostic tests should not have a high rate of "false positives" and also because this increases the time and costs needed to complete diagnostic investigation in patients with defecatory disorders.

The high rate of abnormal findings in healthy individuals may be because current manometry procedures and other anorectal tests (e.g. rectal balloon expulsion) are usually performed, not in the upright, seated position (USP) usually adopted for defecation, but in the un-physiological left lateral position (LLP). Several factors may contribute. First, defecation in the LLP is not aided by gravity as it is in the sitting position. Second, anorectal anatomy may be altered and less conducive to the passage of stool in the LLP. Third, simulating defecation in the LLP does not reflect normal behavior and, despite optimal interaction and explanation by the investigator, changes in patient behavior may result in apparent "dyssynergia" Finally, social stress, related to proximity of the investigator observing defecation, makes individuals feel unable to strain at stool or attempt defecation.

A simple probe holder device that, by adhering to the skin is positioned at the natal cleft to support the ManoScan HR ARM catheter can be used to assess anorectal pressures in the sitting position (both produced by Given Imaging, Yoqeam, Israel). This simple device stabilizes the catheter position when the patient is in USP on a commode and allows the investigator to withdraw behind the curtains of the examination cubicle.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria: All

* Signed informed consent
* Male or female, age 18 - 75 years
* Females eligible to participate either if physiologically incapable of becoming pregnant or with a negative urine pregnancy test at screening
* HS: Absence of symptoms of constipation or incontinence

Patients with fecal incontinence

* Passive or Urge Incontinence
* Wexner Score of 5-20 ("more than mild severity of incontinence")

Patients with obstructive defecation

• Cleveland Clinic Constipation Scoring System: 10-30 ("more than mild severity of constipation)

Exclusion Criteria:

* • Participation in any other clinical trial with investigational or approved drugs within the last month before the study

  * Significant medical, surgical or psychiatric disease requiring on-going active management
  * Previous gastrointestinal or gynaecological disease (exception: non symptomatic ovarian cysts, occasional reflux, appendectomy, hysterectomy, cholecystectomy)
  * Regular use of opiates or other constipating agents
  * Presence of fecal impaction on clinical per rectal exam
  * Abnormal findings on proctoscopy / endoscopy (e.g. Inflammatory Bowel Disease, neoplasm, acute or chronic anal fissure, large haemorrhoids (grade 3-4) intussusception, prolapse or gross perineal descent (>5cm) on straining
  * Insufficient understanding of German language to comply with instructions
  * Contraindication for MRI: Presence of non-MR-compatible metallic implants, devices or metallic foreign bodies

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Recto-anal pressure gradient (RAPG) | 1 hour
  RAPG change in the LLP and sitting position (mmHg)

SECONDARY OUTCOMES:
Presence of dyssynergia on HR-ARM | 1 hour
  RAPG of -40mmHg or lower
Presence of dyssynergic defecation on MRI in healthy controls | 1 hour
  paradox contraction or no opening of the anal canal
Agreement of MR findings in different body positions with HR-ARM findings | 1 hour
  diagnostic concordance of the two investigations
Patient positional preference | 1 hour
  Categorical (forced choice) LLP vs. SEAT

CONTACTS AND LOCATIONS:
Overall Officials: Henriette Heinrich, Study Director — Department for Gastroenterology and Hepatology
Locations (1):
- Department for Gastroenterology and Hepatology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Bharucha AE, Pemberton JH, Locke GR 3rd. American Gastroenterological Association technical review on constipation. Gastroenterology. 2013 Jan;144(1):218-38. doi: 10.1053/j.gastro.2012.10.028. No abstract available. PMID 23261065
- [Background] Ratuapli SK, Bharucha AE, Noelting J, Harvey DM, Zinsmeister AR. Phenotypic identification and classification of functional defecatory disorders using high-resolution anorectal manometry. Gastroenterology. 2013 Feb;144(2):314-322.e2. doi: 10.1053/j.gastro.2012.10.049. Epub 2012 Nov 7. PMID 23142135
- [Background] Noelting J, Ratuapli SK, Bharucha AE, Harvey DM, Ravi K, Zinsmeister AR. Normal values for high-resolution anorectal manometry in healthy women: effects of age and significance of rectoanal gradient. Am J Gastroenterol. 2012 Oct;107(10):1530-6. doi: 10.1038/ajg.2012.221. Epub 2012 Sep 18. PMID 22986439
- [Background] Heinrich H, Fruehauf H, Sauter M, Steingotter A, Fried M, Schwizer W, Fox M. The effect of standard compared to enhanced instruction and verbal feedback on anorectal manometry measurements. Neurogastroenterol Motil. 2013 Mar;25(3):230-7, e163. doi: 10.1111/nmo.12038. Epub 2012 Nov 6. PMID 23130678